CLINICAL TRIAL: NCT05454254
Title: Effect of Muscle Strengthening Training in Adults with Fontan Circulation Compared to Healthy Controls
Brief Title: Effect of Muscle Strengthening Training in Adults with Fontan Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Muscle training Fontan
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease; Univentricular Heart
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adults with Fontan circulation (Active Comparator): Individualised muscle strengthening exercise training protocol.
  Interventions: Other: Individualised muscle strengthening exercise training protocol.
- Healthy controls (Active Comparator): Individualised muscle strengthening exercise training protocol.
  Interventions: Other: Individualised muscle strengthening exercise training protocol.

INTERVENTIONS:
Other: Individualised muscle strengthening exercise training protocol. — Based on the results of muscle function tests at baseline an individualised exercise protocol will be designed.

SUMMARY:
Aim: to evaluate the effect of muscle strengthening exercise training in adults with Fontan circulation compared to healthy controls.

Hypothesis: adults with Fontan circulation have a relatively lower effect of muscle strengthening exercise training compared to healthy controls.

DETAILED DESCRIPTION:
10 adults with Fontan circulation will be recruited from the clinic specialised in adults with congenital heart disease at Norrlands Universitetssjukhus. In addition, 10 age- and sex matched controls will be recruited. The sample size is estimated according to a previous study with the same primary outcome. We estimate that 7 patients and 7 controls are needed in the study and plan to enrol 10 patients and 10 controls in case of any drop outs.

Muscle tests will be performed at baseline. Based on the results from the muscle tests, an individualised muscle training exercise protocol will be designed and the participants will be working out at a gym during 10 weeks. After 10 weeks the same tests will be performed to evaluate the effect of the muscle training exercise.

In addition to the muscle tests, muscle mass and aerobic exercise capacity will be evaluated with peripheral quantitative computed tomography and cardiopulmonary exercise test respectively. Physical activity will be mapped with a validated questionnaire (IPAQ) and an accelerometer attached to the participants thigh. Any impact on fatigue will be evaluated with a validated questionnaire (MFI-20). All tests and questionnaires will be performed at baseline and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum 18 years
* Patients: Congenital heart disease (Fontan circulation, univentricle heart)
* Controls: no known congenital heart disease.

Exclusion Criteria:

* Muscle strenghtening exercise training at regular basis (2 times/week or more)
* Active disease or other condition that affect exercise training (e.g. rheumatoid arthritis)
* Cognitive or psychological affection
* Other conditions that affect independent decision-making competence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle oxygenation kinetics evaluated with near-infrared spectroscopy (NIRS). | 10 weeks
  Muscle oxygenation kinetics will be evaluated with near-infrared spectroscopy (NIRS) (PortaLite mini, Artinis medical system BV, Netherlands). With light in the near infrared spectra it is possible to measure oxygenated and deoxygenated haemoglobin within the muscle. the muscle oxygenation kinetics till be evaluated pre, during and post exercise of muscle endurance in shoulder flexion and heel raise.

SECONDARY OUTCOMES:
Change of isometric muscle strength | 10 weeks
  Isometric muscle strength in elbow flexion and knee extension will be assessed with a load cell amplifier (VZ101BH 500kg, Anyload Weigh & Measure Inc.,NJ, US). Maximal muscle contraction will be performed during five seconds. The test is repeated three times with a one-minute rest in between. Isometric grip strength will be assessed with a handheld dynamometer (JAMAR, Lafayette, IN, USA). The handle is pressed during three seconds and the test is repeated three times, with a one-minute rest in between. The tests are performed at baseline and at follow up after 10 weeks muscle training exercise protocol.
Change of muscular endurance | 10 weeks
  Muscle endurance in shoulder flexion will be assessed with a dumbbell (women 2 kg, men 3 kg) and performed in pace with a metronome, 20 contractions per minute (40 beats per minute). Muscle endurance in the calf muscles will be assessed with heel raise with 10 degrees dorsal flexion in the ankle. The test is performed in pace with a metronome with 30 contractions per minute (60 beats per minute). To evaluate muscle endurance in elbow flexion and knee extension, the test person lifts a weight representing 80% of repetition maximum measured at isometric strength. During all tests, the test person performs as many contractions as possible.
Change of muscle mass | 10 weeks
  Evaluation of muscle mass and muscle density is performed with peripheral quantitative computed tomography (PQCT) which analyse cross section of under arms and lower legs with a low radiation dose (0.01 mSV).
Change of aerobic exercise capacity | 10 weeks
  Cardiopulmonary exercise tests (CPET) are performed according to standardised protocols with incremental increase of workload. During CPET oxygen and carbon dioxide is measured continuously in the inhaled and exhaled air. Peak watt and peak oxygen uptake capacity (peak VO2) is noted. CPET is used to evaluate the effect of muscle strengthening exercise on the aerobic capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wikner A, Rinnstrom D, Johansson K, Bergman F, Ljungberg J, Johansson B, Sandberg C. Positive effects of strength training on dynamic muscle function in adults with Fontan circulation: a pilot study. Cardiol Young. 2025 Dec 22:1-8. doi: 10.1017/S1047951125110457. Online ahead of print. PMID 41424146